CLINICAL TRIAL: NCT03022422
Title: Protective Mechanisms Against a Pandemic Respiratory Virus: B-Cell, T-cell, and General Immune Response to Seasonal Influenza Vaccine. Year 3, 2011
Brief Title: T-cell And General Immune Response to Seasonal Influenza Vaccine (SLVP018) Year 3, 2011
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-17219-2011; 2U19AI057229-06 (NIH)
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Influenza
Keywords: Trivalent, inactivated influenza vaccine; High-Dose trivalent, inactivated influenza vaccine; Adult and elderly identical twins; Adult fraternal twins
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (6):
- Group B: 18-30 yo identical twins (TIV) (Other): Individual twins to receive Fluzone® standard TIV
  Interventions: Biological: TIV
- Group C: 18-30 yo fraternal twins (TIV) (Other): Individual twins to receive Fluzone® standard TIV
  Interventions: Biological: TIV
- Group D: 40-64 yo identical twins (TIV) (Other): Individual twins to receive Fluzone® standard TIV
  Interventions: Biological: TIV
- Group E: 40-64 yo fraternal twins (TIV) (Other): Individual twins to receive Fluzone® standard TIV
  Interventions: Biological: TIV
- Group F: 65-100 yo identical twins (TIV) (Other): Individual twins to receive Fluzone® standard TIV
  Interventions: Biological: TIV
- Group F: 65-100 yo identical twins (High-Dose TIV) (Other): Individual twins to receive High-Dose Fluzone® TIV
  Interventions: Biological: High-Dose TIV

INTERVENTIONS:
Biological: TIV — Influenza Virus Vaccine Suspension for Intramuscular Injection
  Other Names: Fluzone® TIV
  Arms: Group B: 18-30 yo identical twins (TIV); Group C: 18-30 yo fraternal twins (TIV); Group D: 40-64 yo identical twins (TIV); Group E: 40-64 yo fraternal twins (TIV); Group F: 65-100 yo identical twins (TIV)
Biological: High-Dose TIV — High-Dose Influenza Virus Vaccine supplied in a prefilled, single-dose syringe for intramuscular injection
  Other Names: High-Dose Fluzone® TIV
  Arms: Group F: 65-100 yo identical twins (High-Dose TIV)

SUMMARY:
This study will investigate markers, mechanisms and define general predictors for immunological health by comparing influenza vaccine responses in monozygotic and dizygotic twins.

DETAILED DESCRIPTION:
The investigators plan to study the response to influenza vaccines much more broadly and deeply across different age groups and with different vaccine formulations and to probe the influence of genetics on these responses using monozygotic and dizygotic twins. On an investigational basis, investigators plan to compare various immunological responses, identify age-specific biomarkers or clusters of markers, quantify the frequency of influenza-specific T-cells pre- and post-vaccination, and determine the effective breadth of T-cell repertoire to an influenza vaccine within an individual as a function of age and to what degree this is genetically determined.

Twin Groups B-E will receive a single administration of the 2011-2012 formulation of seasonal trivalent inactivated influenza vaccine (TIV). Group F, elderly monozygotic twin participants, will be randomly assigned to receive a single dose of inactivated vaccine, either the usual dose or the High-Dose TIV. Blood samples to conduct the assays described will be taken at pre-immunization, Days 7-10 and 28 post-immunization. The number of individual participants, not the number of twin pairs is being reported in all the modules.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy, ambulatory adults, ages 18-30 years (identical or fraternal twin pairs), 40-64 years (identical or fraternal twin pairs) or 65-100 years (identical twin pairs).
2. Willing to complete the informed consent process.
3. Availability for follow-up for the planned duration of the study at least 28 days after immunization.
4. Acceptable medical history and vital signs.

Exclusion Criteria:

1. Prior off-study vaccination with trivalent inactivated influenza vaccine (TIV) or live attenuated influenza vaccine (LAIV) in Fall 2011
2. Allergy to egg or egg products, or to vaccine components, including thimerosal (if TIV multidose vials used)
3. Allergy to latex (for Group F only - may be assigned to Fluzone High-Dose). Review with investigator.
4. Life-threatening reactions to previous influenza vaccinations
5. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
6. History of immunodeficiency (including HIV infection)
7. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
8. Blood pressure >150 systolic or > 95 diastolic at Visit 1
9. Hospitalization in the past year for congestive heart failure or emphysema.
10. Chronic Hepatitis B or C
11. Recent or current use of immunosuppressive medication, including glucocorticoids (corticosteroid nasal sprays, topical steroids and inhaled steroids are permissible). Use of oral steroids (<20mg prednisone-equivalent/day) may be acceptable after review by the investigator.
12. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
13. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
14. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
15. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except aspirin up to 325 mg.day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
16. Receipt of blood or blood products within the past 6 months
17. Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
18. Inactivated vaccine 14 days prior to vaccination
19. Live, attenuated vaccine within 60 days of vaccination
20. History of Guillain-Barre Syndrome
21. Pregnant or lactating woman
22. Use of investigational agents within 30 days prior to enrollment
23. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment
24. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Dekker, MD, Principal Investigator — Stanford University; Mark Davis, PhD, Principal Investigator — Stanford University; Garry Nolan, PhD, Principal Investigator — Stanford University; Ann Arvin, MD, Principal Investigator — Stanford University; Stephen Quake, PhD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kay AW, Fukuyama J, Aziz N, Dekker CL, Mackey S, Swan GE, Davis MM, Holmes S, Blish CA. Enhanced natural killer-cell and T-cell responses to influenza A virus during pregnancy. Proc Natl Acad Sci U S A. 2014 Oct 7;111(40):14506-11. doi: 10.1073/pnas.1416569111. Epub 2014 Sep 22. PMID 25246558
- [Background] O'Gorman WE, Huang H, Wei YL, Davis KL, Leipold MD, Bendall SC, Kidd BA, Dekker CL, Maecker HT, Chien YH, Davis MM. The Split Virus Influenza Vaccine rapidly activates immune cells through Fcgamma receptors. Vaccine. 2014 Oct 14;32(45):5989-97. doi: 10.1016/j.vaccine.2014.07.115. Epub 2014 Sep 6. PMID 25203448
- [Background] Brodin P, Jojic V, Gao T, Bhattacharya S, Angel CJ, Furman D, Shen-Orr S, Dekker CL, Swan GE, Butte AJ, Maecker HT, Davis MM. Variation in the human immune system is largely driven by non-heritable influences. Cell. 2015 Jan 15;160(1-2):37-47. doi: 10.1016/j.cell.2014.12.020. PMID 25594173
- [Derived] Cheung P, Vallania F, Warsinske HC, Donato M, Schaffert S, Chang SE, Dvorak M, Dekker CL, Davis MM, Utz PJ, Khatri P, Kuo AJ. Single-Cell Chromatin Modification Profiling Reveals Increased Epigenetic Variations with Aging. Cell. 2018 May 31;173(6):1385-1397.e14. doi: 10.1016/j.cell.2018.03.079. Epub 2018 Apr 26. PMID 29706550
- [Derived] de Bourcy CFA, Dekker CL, Davis MM, Nicolls MR, Quake SR. Dynamics of the human antibody repertoire after B cell depletion in systemic sclerosis. Sci Immunol. 2017 Sep 29;2(15):eaan8289. doi: 10.1126/sciimmunol.aan8289. PMID 28963118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Numbers listed in the tables reflect individual twins and not twin pairs.
Groups:
- Group B: 18-30 yo Identical Twins (TIV); Group C: 18-30 yo Fraternal Twins (TIV); Group D: 40-64 yo Identical Twins (TIV); Group E: 40-64 yo Fraternal Twins (TIV): Individual Twins to receive Fluzone® standard TIV
  Fluzone® standard TIV: Influenza Virus Vaccine Suspension for Intramuscular Injection
- Group F: 65-100 yo Identical Twins (TIV): Individual Twins will receive Fluzone® standard TIV: Influenza Virus Vaccine Suspension for Intramuscular Injection
- Group F: 65-100 yo Identical Twins (High-Dose TIV): Individual Twins will receive High-Dose Fluzone® TIV: High-Dose Influenza Virus Vaccine supplied in a prefilled, single-dose syringe for Intramuscular Injection
Period: Overall Study
Arm/Group | Group B: 18-30 yo Identical Twins (TIV) | Group C: 18-30 yo Fraternal Twins (TIV) | Group D: 40-64 yo Identical Twins (TIV) | Group E: 40-64 yo Fraternal Twins (TIV) | Group F: 65-100 yo Identical Twins (TIV) | Group F: 65-100 yo Identical Twins (High-Dose TIV)
Started | 8 | 10 | 23 | 12 | 5 | 5
Completed | 8 | 10 | 20 | 12 | 5 | 5
Not Completed | 0 | 0 | 3 | 0 | 0 | 0
Not completed — 3 subjects consented but not vaccinated | 0 | 0 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Numbers listed in the tables reflect individual twins and not twin pairs. In Group D, one twin of an identical pair consented but was not eligible, so this participant did not receive vaccine. Because of this, the other twin of this identical pair did not come in for a study visit.
Groups:
- Group F: 65-100 yo Identical Twins (High-DoseTIV): Individual twins will receive Fluzone® high-dose TIV: High-Dose Influenza Virus Vaccine supplied in a prefilled, single-dose syringe for Intramuscular Injection
- Total: Total of all reporting groups
Arm/Group | Group B: 18-30 yo Identical Twins (TIV) | Group C: 18-30 yo Fraternal Twins (TIV) | Group D: 40-64 yo Identical Twins (TIV) | Group E: 40-64 yo Fraternal Twins (TIV) | Group F: 65-100 yo Identical Twins (TIV) | Group F: 65-100 yo Identical Twins (High-DoseTIV) | Total
Number analyzed (Participants) | 8 | 10 | 23 | 12 | 5 | 5 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.79 (4.18) | 26.37 (3.11) | 50.55 (7.03) | 55.86 (7.10) | 70.08 (3.83) | 70.08 (3.83) | 47.55 (16.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 15 | 7 | 3 | 3 | 42
  Male | 2 | 2 | 8 | 5 | 2 | 2 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity is reported as self-identified; identical twins could have provided different responses.
  Participants
    Hispanic or Latino | 3 | 1 | 3 | 2 | 0 | 0 | 9
    Not Hispanic or Latino | 5 | 8 | 20 | 10 | 5 | 5 | 53
    Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 8 | 20 | 9 | 5 | 5 | 53
  More than one race | 2 | 2 | 0 | 2 | 0 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 23 | 12 | 5 | 5 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Individual Twins Who Received Influenza Vaccine
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Groups:
- Group F: 65-100 yo Identical Twins (High-DoseTIV): Individual Twins will receive High-Dose Fluzone® TIV: High-Dose Influenza Virus Vaccine supplied in a prefilled, single-dose syringe for Intramuscular Injection
Arm/Group | Group B: 18-30 yo Identical Twins (TIV) | Group C: 18-30 yo Fraternal Twins (TIV) | Group D: 40-64 yo Identical Twins (TIV) | Group E: 40-64 yo Fraternal Twins (TIV) | Group F: 65-100 yo Identical Twins (TIV) | Group F: 65-100 yo Identical Twins (High-DoseTIV)
Number analyzed (Participants) | 8 | 10 | 20 | 12 | 5 | 5
Participants | 8 | 10 | 20 | 12 | 5 | 5

2. Secondary Outcome: Number of Individual Twins With Related Adverse Events
Time Frame: Day 0 to 28 post-immunization
Measure: Count of Participants; unit: Participants
Groups:
- Group F: 65-100 yo Identical Twins (TIV): Individual Twins will receive Fluzone® TIV: Influenza Virus Vaccine Suspension for Intramuscular Injection
Arm/Group | Group B: 18-30 yo Identical Twins (TIV) | Group C: 18-30 yo Fraternal Twins (TIV) | Group D: 40-64 yo Identical Twins (TIV) | Group E: 40-64 yo Fraternal Twins (TIV) | Group F: 65-100 yo Identical Twins (TIV) | Group F: 65-100 yo Identical Twins (High-Dose TIV)
Number analyzed (Participants) | 8 | 10 | 20 | 12 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Group F: 65-100 yo Identical Twins (High-Dose TIV): Participants will receive High-Dose Fluzone® TIV: High-Dose Influenza Virus Vaccine supplied in a prefilled, single-dose syringe for Intramuscular Injection
Arm/Group | Group B: 18-30 yo Identical Twins (TIV) | Group C: 18-30 yo Fraternal Twins (TIV) | Group D: 40-64 yo Identical Twins (TIV) | Group E: 40-64 yo Fraternal Twins (TIV) | Group F: 65-100 yo Identical Twins (TIV) | Group F: 65-100 yo Identical Twins (High-Dose TIV)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10 | 0/20 | 0/12 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/20 | 0/12 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/8 | 1/10 | 1/20 | 0/12 | 0/5 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group B: 18-30 yo Identical Twins (TIV) (N=8) | Group C: 18-30 yo Fraternal Twins (TIV) (N=10) | Group D: 40-64 yo Identical Twins (TIV) (N=20) | Group E: 40-64 yo Fraternal Twins (TIV) (N=12) | Group F: 65-100 yo Identical Twins (TIV) (N=5) | Group F: 65-100 yo Identical Twins (High-Dose TIV) (N=5)
Syncopal episode (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Syncopal episode during phlebotomy at V01
Sialolithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Stone removed from sub-lingual salivary gland.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No